CLINICAL TRIAL: NCT03785834
Title: The Effect of Histopathologic Analysis and Tissue Cultures on Inpatient Management of Cellulitis and Pseudocellulitis
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ben H Kaffenberger, Associate Professor-Clinical Dermatology, Ohio State University
Other Study IDs: 2018H0147
Record Dates: First submitted 2018-12-05; First posted 2018-12-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-01

CONDITIONS: Cellulitis; Pseudocellulitis
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Punch Biopsy — The patient will undergo two 6 mm punch biopsies into the affected extremity at the most proximal portion of the redness.

SUMMARY:
The Investigators wish to study the value of dermatologic testing assessments in differentiating between cellulitis and pseudocellulitis in the inpatient setting. The Investigators propose that by utilizing cutaneous biopsies and tissue cultures in patients that have been admitted to inpatient internal medicine teams, the investigators may be able to improve multiple measures of hospital efficiency in patients presenting with cellulitis-like symptoms, by more accurately recognizing cellulitis from pseudocellulitis. The patient will undergo encrypted digital imaging for his or her condition. This image will then be sent to the study investigators, along with basic clinical information on the skin evaluation form. The study investigators will develop a differential diagnosis and then the patient will undergo a skin biopsy. The patient will then be randomized to one of two arms using a random number generator: A) Skin biopsies and tissue cultures recorded and published in patient's medical chart as they would be in a standard of care procedure B) Skin biopsies and tissue cultures consultation performed but not published in the patient's medical chart unless medically necessary. Information will be collected from medical records in IHIS. Patients will be contacted by phone 30 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* admitted inpatient to The Ohio State University Wexner Medical Center Internal Medicine ward with cellulitis-like symptoms, including but not limited to the following: tenderness, redness, swelling, expansive lesion.
* Affecting one or more extremities
* are at least 90 days post any associated operation of the extremity
* are above the age of 18
* Participants will be patients with cellulitis or pseudocellulitis.
* Patients who have recurrent cellulitis will be eligible for enrollment into the study, but only once.

Exclusion Criteria:

* Patients who are pregnant
* Prisoners
* Patients may not have trauma, ulcer, or puncture wound to the area
* May not be transferred from another hospital
* May not be admitted to the Cancer Hospital or with a known active solid organ or hematologic cancer other than nonmelanoma skin cancer

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's ages 18 to 99 years that present in the ED with pseudocellulitis or cellulitis.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The feasibility of conducting a larger study will be conducted, by establishing patient enrollment rates | At study completion, around 2 years after study start
  According to the NIH: The goal of pilot work is not to test hypotheses about the effects of an intervention, but rather, to assess the feasibility/acceptability of an approach to be used in a larger scale study. We will use descriptive statistics to monitor patient enrollment and pilot data on additional secondary outcomes for inferential statistics.

SECONDARY OUTCOMES:
Change in antibiotic use (antibiotics/day administered) over the course of the hospitalizations | 1 year
  Cellulitis is a common type of bacterial skin infection. Pseudocellulitis is a skin infection that is very similar to cellulitis and is often misdiagnosed as cellulitis
The rate of participant readmission within 30 days | 1 year
  The investigators will examine 30 day readmission rates between standard care and interventional care
Length of hospitalization as measured in days | 1 year
  The investigators will examine hospital length-of-stay in patients randomized to interventional vs standard care

CONTACTS AND LOCATIONS:
Overall Officials: Benhamin Kaffenberger, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Dermatology, Gahanna, Ohio, United States

IPD SHARING:
Plan to Share IPD: No